CLINICAL TRIAL: NCT04267705
Title: Understanding the Pulse-Gut Relationship and it's Role in Modifying Systemic Inflammation and Insulin Sensitivity in Humans
Brief Title: Pulses Consumption and Its Role in Managing Systemic Inflammation, Insulin Sensitivity and Gut Microbiome in Human
Acronym: PS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019-070
Record Dates: First submitted 2020-02-05; First posted 2020-02-13 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Insulin Sensitivity; Overweight or Obesity; Inflammatory Response
Keywords: Pulses; gut microbiota
MeSH Terms: conditions — Insulin Resistance; Overweight; Obesity | interventions — cicerin protein, Cicer arietinum

STUDY DESIGN:
Intervention Model Description: The proposed study is a randomized, 3-arm, parallel, placebo-controlled design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Black bean (Active Comparator): A cup of black bean 7 days/week over a 12-week period
  Interventions: Other: Black bean
- Chickpea (Active Comparator): A cup of chickpea 7 days/week over a 12-week period
  Interventions: Other: Chickpea
- Control (Placebo Comparator): A cup of white rice 7 days/week over a 12-week period
  Interventions: Other: Control

INTERVENTIONS:
Other: Control — This group will receive a cup of rice 7 days/week over a 12-week period
  Arms: Control
Other: Black bean — This group will receive a cup of black bean7 days/week over a 12-week period
  Arms: Black bean
Other: Chickpea — This group will receive a cup of chick pea 7 days/week over a 12-week period
  Arms: Chickpea

SUMMARY:
Objective 1: Characterize indices of systemic inflammation and gut microbiota composition and function after chronic (12 weeks) intake of pulses compared to control diet in human OW/OB-IR participants.

Objective 2: Characterize dietary- and microbial-derived metabolite pools after regular intake of pulses (12 weeks) in human participants with OW/OB-IR compared to control diet.

Objective 3: Characterize cognitive functioning after chronic (12 weeks) intake of pulses compared to control diet in human OW/OB-IR participants.

DETAILED DESCRIPTION:
The proposed study will be conducted in humans according to Good Clinical Practice (GCP) guidelines. All subjects will review and sign an Informed Consent Form approved by the Illinois Institute of Technology's Institutional Review Boards (IRB) prior to screening.

The proposed study is a randomized, 3-arm, parallel, placebo-controlled design to investigate the effects of pulses consumption compared to non-pulse foods on indices of systemic inflammation and gut microbiota composition and function over a 12-week period. Potential changes in cognition will also be assessed. The study will test 3 treatment conditions in overweight (OW)/obese (OB) human subjects with insulin resistant (IR). Eighty-three men and women will be recruited, aiming for a completer set of Sixty-six subjects. Participants will be randomized into one of the three study food intervention groups:

1. Control group, (n=22): This group will receive a cup of white rice 7 days/week over a 12-week period.
2. Black bean group, (n=22): This group will receive a cup of black bean 7 days/week over a 12-week period.
3. Chickpea group, (n=22): This group will receive a cup of chickpea 7 days/week over a 12-week period.

Each subject will be asked to come for 1 Screening Visit, 4 biweekly food pick-up/compliance visits and 3 Test Day Visits (two of which will also include cognitive testing). The initial screening visit will provide subjects with their site-specific, IRB-approved informed consent document prior to the start of any study-related procedures. Following 1-week diet stabilization and wash in from anthocyanins and ellagitannins, eligible subjects will be randomized to receive 1 of 3 test treatments based on a randomization schedule. The three main Test Day visits will occur at week 0 (day 1; baseline), end of week 6 (mid-point) and at the end of week 12 (end-point). Cognitive testing will occur during the baseline Test Day at week 0, and again at end-point Test Day at week 12. Subjects will be given a breakfast meal before cognitive testing. Pick-up Visits will occur at week 2, 4, 8, and 10. Subjects will pick-up study foods receive dietary counseling, confirm diet compliance and have anthropometrics checked during pick-up visits. Each of the 3 Test Day Visits will last about 2.5-3 h (not including cognitive testing) and involve blood pressure (BP) measurements, anthropometric (weight, waist circumference; body composition) assessment, and an oral glucose tolerance test (OGTT) will be performed. Urine and fecal samples will be collected to monitor modifications occurring in the metabolites during the supplementation. The two-Test Day Visits (baseline and end-point) will also include an additional 1-1.25 h of cognitive testing, for a total of 3.75-4.5 h of total subject time (as there will be a short break between OGTT and cognitive testing). Subjects will maintain daily food and GI-tract diary during the 12-week feeding trial. The diary will include questions about food intake and the condition of gastrointestinal tolerance and bowel function.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, age 18 or older
* BMI ≥ 25 kg/m2
* Fasting blood glucose concentration between 100 mg/dL and 125 mg/dL at the screening visit
* Nonsmokers (Past smokers can be allowed if they have abstinence for a minimum of 2 years)
* Judged to be in good health on the basis of the medical history ie., no clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
* Not taking any medications that would interfere with outcomes of the study, i.e. lipid-lowering medications, anti-inflammatory drugs, dietary supplements, etc.
* Able to provide informed consent
* Able to comply and perform the procedures requested by the protocol (including dietary restrictions, consumption of study treatments, records of food diary and GI-tract questionnaire, sample collection procedures and study visit schedule)
* Able to maintain the usual physical activity pattern
* Able to abstain from alcohol consumption and avoid vigorous physical activity for 24 hours prior to and during the study visit

Exclusion Criteria:

* Men and women who smoke
* Men and women with known or suspected intolerance, allergies or hypersensitivity to study foods or treatments
* Men and women who have blood pressure >160 mmHg (systolic)/100 mmHg (diastolic) at the screening visit
* Men and women who have fasting blood glucose concentration <100 or >125 mg/dL at the screening visit
* Men and women with documented vascular disease, e.g., heart failure, myocardial infarction, stroke, angina, related surgeries, etc. that, in the opinion of the investigator, could interfere with the interpretation of the study results
* Men and women with cancer other than non-melanoma skin cancer in the previous 5 years
* Men and women diagnosed with chronic constipation, diarrhea or other chronic gastrointestinal complaints (e.g. irritable bowel syndrome)
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study
* Women who are lactating
* Taking medication or dietary supplements that may interfere with the outcomes of the study; e.g., antioxidant supplement, anti-inflammation, lipid-lowering medication, blood pressure-lowering medication, etc... Subjects may choose to go off dietary supplements (requires 30 days washout); e.g., fish oil, probiotics, etc...
* Men and women who have participated in prebiotics or laxative trial within 3 months prior to enrollment or any other clinical trial within 1 month
* Major trauma or a surgical event within 2 months or longer depending on trauma or event and after consultation with PI.
* Vegan or other extreme dietary regimens (e.g., Atkins diet, etc.) as judged by the investigator.
* Taking the fiber supplements and/or on high fiber diets
* Has used antibiotics within the previous 2 months
* Had gastrointestinal barium opaque meal within 3 months
* Has used prebiotics, probiotics, or drugs active on gastrointestinal motility, or a laxative of any class within 1 month
* History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional
* Substance (alcohol or drug) abuse within the last 2 years
* Excessive coffee and tea consumers (> 4 cups/d)
* Donated blood within last 3 months
* Men and women who do excessive exercise regularly or are an athlete
* Unstable weight: gained or lost weight +/- 5 kg (11 lbs) in previous 2 months
* Women who are taking unstable dose and brand of hormonal contraceptives and/or stable dose and brand less than 6 months
* Unusual working hours i.e., working overnight (e.g. 3rd shift)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Plasma biomarkers and measures of inflammation: Nrf2/ NF-κB | Baseline to 12 weeks
  Investigate Nrf2/ NF-κB activation in PBMC
Changes in plasma systemic and gut inflammatory markers | Baseline to 12 weeks
  Collected plasma samples will be used to measure selected inflammatory markers (IL6, hs-CRP and TNF-α) using ELISA methods
Determination of GLP-2 in plasma | Baseline to 12 weeks
  Analysis of GLP-2 will be done in plasma samples before and after chronic exposure to the study foods using enzyme Immunoassay (EIA) kit as per manufacturer's instructions.
Determination of TLR-2/4 gene expression in Human PBMC | Baseline to 12 weeks
  Determination of TLR-2/4 gene expression in Human PBMC using RT-PCR method
Gut inflammatory markers: Calprotectin, zonulin, and IgA in fecal samples | Baseline to 12 weeks
  The concentration of calprotectin, zonulin, and IgA in fecal samples will be determined by enzyme-linked immunosorbent assay (ELISA) as per kit providers' instructions before and after chronic exposure to study foods.
Describe functional metagenomics alterations in gut microbiome | Baseline to 12 weeks
  Fecal samples will be collected with standard collection kits and stored at -80°C until analysis. Metagenomic and transcriptomic analyses will be performed

SECONDARY OUTCOMES:
Characterize metabolite profiles | Baseline to 12 weeks
  Polyphenolic metabolites (phenolic acids and derivatives components) will be identified and quantified in urine and plasma.Metabolites in samples will be identified and quantified using an Agilent 6550 iFunnel UHPLC-QTOF-MS and 6460 UHPLC-QQQ-MS, respectively.
Characterize bile acid metabolite pool | Baseline to 12 weeks
  Bile acids in plasma and fecal samples will be determined using UHPLC-QQQ-MS.

OTHER OUTCOMES:
Cognitive assessment: learning | Baseline to 12 weeks
  California Verbal Learning Test® | Second Edition (CVLT®-II) will be measured in baseline and 12 weeks
Cognitive assessment: basic attention, and working memory. | Baseline to 12 weeks
  A subtest of the WAIS-IV, Digit Span will be measured in baseline and 12 weeks
Cognitive assessment: verbal phonemic (letter) and semantic (category) fluency | Baseline to 12 weeks
  Verbal Fluency: FAS + Animals test will be measured in baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Indika Edirisinghe, Ph.D, Principal Investigator — Illinois Insititute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States